CLINICAL TRIAL: NCT04016662
Title: A Randomized Cross-over Trial Evaluating Automated Insulin Delivery Technologies on Hypoglycemia and Quality of Life in Elderly Adults With Type 1 Diabetes
Brief Title: Automated Insulin Delivery in Elderly With Type 1 Diabetes (AIDE T1D)
Acronym: AIDE T1D
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); DexCom, Inc. (Industry); Tandem Diabetes Care, Inc. (Industry); University of Minnesota - Advanced Research and Diagnostic Laboratory (Unknown); Mayo Clinic (Other); University of Pennsylvania (Other); AdventHealth Diabetes Institute (Unknown); Washington State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AIDE T1D
Record Dates: First submitted 2019-07-09; First posted 2019-07-11 (Actual); Results first posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-12

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Randomized crossover trial with three 12-week crossover periods (HCL during one period, PLGS during one period, and SAP therapy (control) during one period) preceded by a run-in phase.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Hybrid Closed Loop Control (HCL) (Active Comparator): The HCL intervention arm will utilize the Tandem t:slim X2 with Control-IQ Technology and Dexcom G6 CGM
  Interventions: Device: Tandem t:slim X2 with HCL or PLGS
- Predictive Low-Glucose Insulin Suspension (PLGS) (Active Comparator): The PLGS intervention arm will utilize the Tandem t:slim X2 with Basal-IQ Technology and Dexcom G6 CGM
  Interventions: Device: Tandem t:slim X2 with HCL or PLGS
- Sensor-Augmented Pump (SAP) (No Intervention): The SAP arm will utilize the Tandem t:slim X2 without HCL or PLGS features turned on and Dexcom G6 CGM

INTERVENTIONS:
Device: Tandem t:slim X2 with HCL or PLGS — The system components include the t:slim X2 with Control-IQ Technology and the Dexcom CGM G6. The modular control algorithm has a safety supervision module that limits insulin delivery to prevent hypoglycemia at all times. The algorithm gradually decreases hyperglycemia from bedtime to reach a target of 120 mg/dL by waking time. During awake hours, the control algorithm attempts to maintain glucose within a target range (112.5 to 160 mg/dL) with meal time insulin boluses delivered based on usual bolus procedures undertaken by patients on an insulin pump (Hybrid closed loop).
  The system components include the t:slim X2 with with Basal-IQ Technology and the Dexcom CGM G6. The PLGS System is able to stop and resume basal insulin delivery automatically in response to predicted or low sensor glucose values, thereby reducing the incidence and duration of hypoglycemic episodes. The pump includes the hypoglycemia minimization strategy that will issue insulin delivery commands.
  Other Names: Tandem t:slim X2 with Control-IQ Technology; Tandem t:slim X2 with Basal-IQ Technology
  Arms: Hybrid Closed Loop Control (HCL); Predictive Low-Glucose Insulin Suspension (PLGS)

SUMMARY:
A multi-center, randomized, crossover trial consisting of three sequential 12-week periods, with the HCL feature used during one period, the PLGS feature used during one period and SAP therapy (control) during one period. The crossover trial will be preceded by a run-in phase in which participants will receive training using the study devices (Dexcom G6 and Tandem t:slim X2 pump). After the last crossover period, participants will be given the opportunity to use study devices for an additional 12 weeks to assess preference of system use (PLGS, HCL or SAP) and associated characteristics, durability and safety in a more real-world setting with less frequent study contact.

DETAILED DESCRIPTION:
Automated insulin delivery (AID) technologies hold the promise of optimizing glycemic control and reducing the burden of diabetes care for patients with Type 1 Diabetes (T1D). However, clinical trials of lower burden AID technologies have not included older adults in sufficient numbers to allow for focused evaluation of efficacy and quality of life (QOL) impacts that may differ from those observed in younger age groups. Most notably, primary endpoints have focused on reducing hyperglycemia, while avoidance of hypoglycemia is of upmost concern for older adults with T1D. T1D Exchange clinic registry data have shown severe hypoglycemia (SH) occurs more commonly in older adults with longstanding T1D than in younger individuals with events occurring just as often with HbA1c levels >8.0% as with HbA1c levels <7.0%. These data do not support the strategy of "raising the HbA1c" as being an effective approach for hypoglycemia prevention in older adults with T1D. In addition to acutely altered mental status, hypoglycemia is associated with an increased risk for falls leading to fractures, car accidents, emergency room (ER) visits, hospitalizations, and mortality resulting in substantial societal costs. The occurrence of hypoglycemia, hypoglycemia unawareness and fear of hypoglycemia have adverse effects on overall QOL of both individuals with T1D and their families.

While continuous glucose monitoring (CGM) technology alone has the potential to be beneficial in reducing hypoglycemia in older patients, our preliminary data from the Wireless Innovations for Seniors with Diabetes Mellitus (WISDM) trial shows a majority of patients still have frequent hypoglycemia even when using CGM. Thus, knowledge of CGM alone may not be sufficient to avoid hypoglycemia in this population. Predictive low-glucose suspend algorithms have particular promise when the primary goal is hypoglycemia avoidance rather than glucose reduction. Whether the added complexity of closed loop systems provides additional glycemic benefit is not known. There is a critical need to determine whether automated insulin delivery can reduce hypoglycemia in the older adult population with T1D.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of type 1 diabetes
2. Age ≥ 65 years old
3. T1D Duration of at least 1 year
4. HbA1c < 10.0% from point of care or local lab within the past 6 months
5. Insulin regimen involves basal/bolus insulin via insulin pump or multiple daily injections
6. Most recent GFR ≥ 30 ml/min/m^2 from local lab within the past 6 months
7. Willingness to use a rapid acting insulin compatible with the Tandem t:slim X2 pump (currently aspart and lispro; other rapid acting insulins likely to be approved for pump use prior to study initiation such as Fiasp)
8. Familiarity with and willingness to use a carbohydrate ratio for meal boluses
9. Willing to use study devices and automated insulin delivery features
10. Ability to download study devices at home or if not able to download at home willing to come into clinic to bring devices for download of data at visits and as needed for safety
11. Participant is independently managing his/her diabetes with respect to insulin administration and glucose monitoring (may include assistance from spouse or other caregiver)
12. Participant understands the study protocol, agrees to comply with it and is able to successfully pass the consent understanding assessment with no more than 2 attempts
13. Participant comprehends written and spoken English
14. At least 240 hours of CGM readings available during the end of run-in assessment
15. At least 1.5% of time with CGM glucose levels < 70 mg/dL prior to SAP initiation
16. Active prescription for glucagon and willing and able to have glucagon available

Exclusion Criteria:

1. Use of PLGS technology or HCL insulin delivery in the past 1 month
2. History of 1 or more Diabetic Ketoacidosis episodes in the previous 6 months
3. Clinical diagnosis by a primary care provider, neurologist or psychiatrist of dementia, in the investigator's opinion a suspected severe cognitive impairment such that it would preclude ability to understand the study or use devices, or a score of 6 or less out of 15 on the 5 min MoCA (5-min T MoCA Version 2.1) (mild cognitive impairment is not an exclusion)
4. A condition, which in the opinion of the investigator or designee, would put the participant or study at risk, including severe vision or hearing impairment and any contraindication to the use of any of the study devices per FDA labeling
5. Known adhesive allergy or skin reaction during the run-in pre-randomization phase or previous difficulty with pump and CGM insertions that would preclude participation in the randomized trial
6. Concurrent use of any non-insulin glucose-lowering agent other than metformin (including GLP-1 agonists, Symlin, DPP-4 inhibitors, SGLT-2 inhibitors, sulfonylureas)
7. Stage 4 or 5 renal disease
8. The presence of a significant medical or psychiatric condition or use of a medication that in the judgment of the investigator may affect completion of any aspect of the protocol, or is likely to be associated with life expectancy of <1 year

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 82 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2024-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Henderson, MS, Principal Investigator — Jaeb Center for Health Research
Locations (4):
- United States (4):
  - AdventHealth Diabetes Institute, Orlando, Florida
  - Mayo Clinic, Rochester, Minnesota
  - SUNY Upstate, Syracuse, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
deidentified data will be shared on the JCHR website
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available after publication of the primary manuscript and will remain available in perpetuity
Access Criteria: users must have a valid email address
URL: https://public.jaeb.org/datasets/diabetes

REFERENCES:
- [Derived] Kudva YC, Henderson RJ, Kanapka LG, Weinstock RS, Rickels MR, Pratley RE, Chaytor N, Janess K, Desjardins D, Pattan V, Peleckis AJ, Casu A, Rizvi SR, Bzdick S, Whitaker KJ, Kamimoto JLJ, Miller K, Kollman C, Beck RW; AIDE Study Group. Automated Insulin Delivery in Elderly with Type 1 Diabetes: A Prespecified Analysis of the Extension Phase. Diabetes Technol Ther. 2025 Jul;27(7):572-575. doi: 10.1089/dia.2024.0560. Epub 2025 Mar 11. PMID 40067490
- [Derived] Kudva YC, Henderson RJ, Kanapka LG, Weinstock RS, Rickels MR, Pratley RE, Chaytor N, Janess K, Desjardins D, Pattan V, Peleckis AJ, Casu A, Rizvi SR, Bzdick S, Whitaker KJ, Jo Kamimoto JL, Miller K, Kollman C, Beck RW. Automated Insulin Delivery in Older Adults with Type 1 Diabetes. NEJM Evid. 2025 Jan;4(1):EVIDoa2400200. doi: 10.1056/EVIDoa2400200. Epub 2024 Dec 23. PMID 39714936

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a crossover study, so the same 82 randomized patients participated in each arm. If they drop out, they might not be in one of the arms.
Groups:
- All Study Participants: All participants were randomized to receive all interventions: Hybrid Closed Loop Control (HCL), Predictive Low-Glucose Insulin Suspension (PLGS), and Sensor-Augmented Pump (SAP).
Period: Run-In Phase
Arm/Group | All Study Participants
Started | 105
Completed | 81
Not Completed | 24
Not completed — Death | 1
Not completed — Withdrawal by Subject | 11
Not completed — Not meeting screening eligibility | 9
Not completed — Physician Decision | 3
Period: HCL (12 Weeks)
Arm/Group | All Study Participants
Started | 81
Completed | 80
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: PLGS (12 Weeks)
Arm/Group | All Study Participants
Started | 80
Completed | 79
Not Completed | 1
Not completed — Death | 1
Period: SAP (12 Weeks)
Arm/Group | All Study Participants
Started | 79
Completed | 78
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: The same 82 patients at baseline participated in each arm unless they dropped or there was a death.
Arm/Group | All Study Participants
Number analyzed (Participants) | 82
Age, Customized [Count of Participants; unit: Participants]
  65-<70 years | 38
  70-<75 years | 33
  75-<80 years | 9
  ≥80 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 82
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 80
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 82
Central Lab Baseline HbA1c (%) [Mean (Standard Deviation); unit: percentage of glycated hemoglobin] | 7.2 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: CGM Measured Time <70 mg/dL
Description: Primary Outcome: Percentage of sensor glucose values <70 mg/dL. The first 4 weeks of CGM data in each period were excluded to reduce the chance of a carryover effect. A minimum of 168 hours of data was required to calculate CGM metrics. Since the hypoglycemia endpoints had skewed distributions, values were winsorized at the 10th and 90th percentiles.
Time Frame: weeks 5-12 of 12 weeks for each intervention of the crossover
Measure: Mean (Standard Deviation); unit: % time <70 mg/dL
Groups:
- Hybrid Closed Loop Control (HCL): The HCL intervention arm will utilize the Tandem t:slim X2 with Control-IQ Technology and Dexcom G6 CGM
  Tandem t:slim X2 with HCL or PLGS: The system components include the t:slim X2 with Control-IQ Technology and the Dexcom CGM G6. The modular control algorithm has a safety supervision module that limits insulin delivery to prevent hypoglycemia at all times. The algorithm gradually decreases hyperglycemia from bedtime to reach a target of 120 mg/dL by waking time. During awake hours, the control algorithm attempts to maintain glucose within a target range (112.5 to 160 mg/dL) with meal time insulin boluses delivered based on usual bolus procedures undertaken by patients on an insulin pump (Hybrid closed loop).
  The system components include the t:slim X2 with with Basal-IQ Technology and the Dexcom CGM G6. The PLGS System is able to stop and resume basal insulin delivery automatically in response to predicted or low sensor glucose values, thereby reducing the incidence and duration of hypoglycemic episodes. The pump includes the hypoglycemia minimization strategy that will issue insulin delivery commands.
- Predictive Low-Glucose Insulin Suspension (PLGS): The PLGS intervention arm will utilize the Tandem t:slim X2 with Basal-IQ Technology and Dexcom G6 CGM
  Tandem t:slim X2 with HCL or PLGS: The system components include the t:slim X2 with Control-IQ Technology and the Dexcom CGM G6. The modular control algorithm has a safety supervision module that limits insulin delivery to prevent hypoglycemia at all times. The algorithm gradually decreases hyperglycemia from bedtime to reach a target of 120 mg/dL by waking time. During awake hours, the control algorithm attempts to maintain glucose within a target range (112.5 to 160 mg/dL) with meal time insulin boluses delivered based on usual bolus procedures undertaken by patients on an insulin pump (Hybrid closed loop).
  The system components include the t:slim X2 with with Basal-IQ Technology and the Dexcom CGM G6. The PLGS System is able to stop and resume basal insulin delivery automatically in response to predicted or low sensor glucose values, thereby reducing the incidence and duration of hypoglycemic episodes. The pump includes the hypoglycemia minimization strategy that will issue insulin delivery commands.
Arm/Group | Hybrid Closed Loop Control (HCL) | Predictive Low-Glucose Insulin Suspension (PLGS) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 81 | 79 | 78
% time <70 mg/dL | 1.58 (0.95) | 1.67 (0.96) | 2.57 (1.54)

2. Secondary Outcome: CGM Measured Time <54 mg/dL
Description: Percentage of sensor glucose values <54 mg/dL. The first 4 weeks of CGM data in each period were excluded to reduce the chance of a carryover effect. A minimum of 168 hours of data was required to calculate CGM metrics. Since the hypoglycemia endpoints had skewed distributions, values were winsorized at the 10th and 90th percentiles.
Time Frame: weeks 5-12 of 12 weeks for each intervention of the crossover
Measure: Mean (Standard Deviation); unit: % time <54 mg/dL
Arm/Group | Hybrid Closed Loop Control (HCL) | Predictive Low-Glucose Insulin Suspension (PLGS) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 81 | 79 | 78
% time <54 mg/dL | 0.29 (0.23) | 0.27 (0.20) | 0.48 (0.40)

3. Secondary Outcome: Hypoglycemia
Description: Rate of CGM-measured hypoglycemic events per week. A hypoglycemic event is defined as 15 consecutive minutes with a sensor glucose value <54 mg/dl. At least 2 sensor values <54 mg/dl that are 15 or more minutes apart plus no intervening values >54 mg/dl are required to define an event. The end of the hypoglycemic event is defined as a minimum of 15 consecutive minutes with a sensor glucose concentration >70 mg/dl. At least 2 sensor values >70 mg/dl that are 15 or more minutes apart with no intervening values <70 mg/dl, are required to define the end of an event. When a hypoglycemic event ends, the study participant becomes eligible for a new event.
Time Frame: weeks 5-12 of 12 weeks for each arm of the crossover
Measure: Mean (Standard Deviation); unit: hypoglycemic events per week
Arm/Group | Hybrid Closed Loop Control (HCL) | Predictive Low-Glucose Insulin Suspension (PLGS) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 81 | 79 | 78
hypoglycemic events per week | 0.6 (0.5) | 0.5 (0.5) | 0.9 (0.8)

4. Secondary Outcome: Glucose Control
Description: Mean glucose (mg/dL)
Time Frame: weeks 5-12 of 12 weeks for each arm of the crossover
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Hybrid Closed Loop Control (HCL) | Predictive Low-Glucose Insulin Suspension (PLGS) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 81 | 79 | 78
mg/dL | 152 (16) | 161 (23) | 160 (20)

5. Secondary Outcome: % Time 70-180 mg/dL
Description: Percentage of sensor glucose values 70 to 180 mg/dL. The first 4 weeks of CGM data in each period were excluded to reduce the chance of a carryover effect. A minimum of 168 hours of data was required to calculate CGM metrics.
Time Frame: weeks 5-12 of 12 weeks for each intervention of the crossover
Measure: Mean (Standard Deviation); unit: % time in range 70-180 mg/dL
Arm/Group | Hybrid Closed Loop Control (HCL) | Predictive Low-Glucose Insulin Suspension (PLGS) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 81 | 79 | 78
% time in range 70-180 mg/dL | 74 (10) | 67 (14) | 66 (12)

6. Secondary Outcome: Glucose Control - Coefficient of Variation
Description: Coefficient of variation (%)
Time Frame: weeks 5-12 of 12 weeks for each arm of the crossover
Measure: Mean (Standard Deviation); unit: % coefficient of variation
Arm/Group | Hybrid Closed Loop Control (HCL) | Predictive Low-Glucose Insulin Suspension (PLGS) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 81 | 79 | 78
% coefficient of variation | 33 (5) | 35 (4) | 36 (5)

7. Secondary Outcome: % Time > 180 mg/dL
Description: Percentage of values >180 mg/dL. The first 4 weeks of CGM data in each period were excluded to reduce the chance of a carryover effect. A minimum of 168 hours of data was required to calculate CGM metrics.
Time Frame: weeks 5-12 of 12 weeks for each intervention of the crossover
Measure: Mean (Standard Deviation); unit: % of time >180 mg/dL
Arm/Group | Hybrid Closed Loop Control (HCL) | Predictive Low-Glucose Insulin Suspension (PLGS) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 81 | 79 | 78
% of time >180 mg/dL | 24 (10) | 31 (14) | 31 (13)

8. Secondary Outcome: % Time > 250 mg/dL
Description: Percentage of values >250 mg/dL. The first 4 weeks of CGM data in each period were excluded to reduce the chance of a carryover effect. A minimum of 168 hours of data was required to calculate CGM metrics.
Time Frame: weeks 5-12 of 12 weeks for each intervention of the crossover
Measure: Mean (Standard Deviation); unit: % of time >250 mg/dL
Arm/Group | Hybrid Closed Loop Control (HCL) | Predictive Low-Glucose Insulin Suspension (PLGS) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 81 | 79 | 78
% of time >250 mg/dL | 5.6 (5.2) | 8.7 (8.8) | 8.6 (7.0)

9. Secondary Outcome: HbA1c
Description: HbA1c %
Time Frame: at 12 week visit for each arm of the crossover
Measure: Mean (Standard Deviation); unit: % of HbA1c
Arm/Group | Hybrid Closed Loop Control (HCL) | Predictive Low-Glucose Insulin Suspension (PLGS) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 75 | 73 | 70
% of HbA1c | 6.9 (0.7) | 7.1 (0.8) | 7.0 (0.8)

10. Secondary Outcome: Hypoglycemia Unawareness - Gold Survey
Description: The Gold score asks subjects to indicate their awareness of hypoglycemia with '1' being always aware and '7' being never aware.
  Score scale 1-7; A higher score indicates more unawareness.
Time Frame: at 12 week visit for each arm of the crossover
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hybrid Closed Loop Control (HCL) | Predictive Low-Glucose Insulin Suspension (PLGS) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 78 | 79 | 76
score on a scale | 2.6 (1.6) | 2.7 (1.5) | 2.9 (1.9)

11. Other Pre Specified Outcome: Patient Reported Questionnaires - Hypoglycemia Fear Survey
Description: The Hypoglycemia Fear Survey measures several dimensions of fear of hypoglycemia among adults with type 1 diabetes. It consists of a 15-item Behavior subscale that measures behaviors involved in avoidance and over-treatment of hypoglycemia and a 18-item Worry subscale that measures anxiety and fear surrounding hypoglycemia. Scores will be calculated overall and for the worry subscale.
  Score scale 0-4; A higher score indicates more fear.
Time Frame: at 12 week visit for each arm of the crossover
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hybrid Closed Loop Control (HCL) | Predictive Low-Glucose Insulin Suspension (PLGS) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 68 | 69 | 64
score on a scale | 0.9 (0.6) | 1.0 (0.6) | 1.0 (0.6)

12. Other Pre Specified Outcome: Patient Reported Questionnaires - Hypoglycemia Confidence
Description: The HCS is a 9-item scale that examines the degree to which people with diabetes feel able, secure, and comfortable regarding their ability to stay safe from hypoglycemic-related problems.
  Score scale 1-4.; A higher score indicates more confidence.
Time Frame: at 12 week visit for each arm of the crossover
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hybrid Closed Loop Control (HCL) | Predictive Low-Glucose Insulin Suspension (PLGS) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 68 | 69 | 64
score on a scale | 3.4 (0.5) | 3.4 (0.5) | 3.4 (0.5)

13. Other Pre Specified Outcome: Patient Reported Questionnaires - Diabetes Distress Scale
Description: 28-item questionnaire used to measure diabetes-related concerns about powerlessness, management, hypoglycemia, social perceptions, eating, physician, and friends/family.
  Score scale 1-6; A higher score indicates more distress.
Time Frame: at 12 week visit for each arm of the crossover
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hybrid Closed Loop Control (HCL) | Predictive Low-Glucose Insulin Suspension (PLGS) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 68 | 69 | 64
score on a scale | 1.6 (0.5) | 1.7 (0.5) | 1.6 (0.6)

14. Other Pre Specified Outcome: Patient Reported Questionnaires - AIDE Technology Acceptance
Description: This diabetes technology specific questionnaire based on the Technology Acceptance Model, assesses perceived system usefulness, ease of use and trust in the system.
  Score scale 1-5; A higher score indicates a more positive appraisal of the system.
Time Frame: at 12 week visit for each arm of the crossover
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hybrid Closed Loop Control (HCL) | Predictive Low-Glucose Insulin Suspension (PLGS) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 68 | 68 | 63
score on a scale | 4.1 (0.6) | 4.0 (0.7) | 3.9 (0.8)

15. Other Pre Specified Outcome: Patient Reported Questionnaires - System Usability
Description: A 10-item questionnaire that measures overall perceived usability of a system and is technology-agnostic.
  Score scale 0-100; Higher score indicates better usability
Time Frame: at 12 week visit for each arm of the crossover
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hybrid Closed Loop Control (HCL) | Predictive Low-Glucose Insulin Suspension (PLGS) | Sensor-Augmented Pump (SAP)
Number analyzed (Participants) | 68 | 69 | 64
score on a scale | 77 (17) | 76 (17) | 73 (16)

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the entirety of the study for the participant (e.g. ~54 weeks)
Groups:
- Run-In Phase: Run-In Phase precedes the randomized assigned treatment groups and includes the CGM Training Period, SAP Training Period, and SAP Evaluation. Length of run-in phase varied depending on participant's prior experience with devices.
Arm/Group | Run-In Phase | Hybrid Closed Loop Control (HCL) | Predictive Low-Glucose Insulin Suspension (PLGS) | Sensor-Augmented Pump (SAP)
All-Cause Mortality (participants affected / at risk) | 1/105 | 0/81 | 1/80 | 1/79
Serious Adverse Events (participants affected / at risk) | 2/105 | 8/81 | 3/79 | 3/78
Other Adverse Events (participants affected / at risk) | 7/105 | 4/81 | 16/79 | 10/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Run-In Phase (N=105) | Hybrid Closed Loop Control (HCL) (N=81) | Predictive Low-Glucose Insulin Suspension (PLGS) (N=79) | Sensor-Augmented Pump (SAP) (N=78)
Diabetic ketoacidosis (Blood and lymphatic system disorders) | 1 | 2 | 0 | 0
Hypoglycemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 2
Hyperglycemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Osteomyelitis (General disorders) | 0 | 1 | 0 | 0
Severe hypoglycemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1
Fluid overload (General disorders) | 0 | 1 | 0 | 0
Ketosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Peripheral arterial disease (General disorders) | 0 | 0 | 1 | 0 — The participant was admitted to the hospital for an elective procedure
Intracranial hemorrhage (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Run-In Phase (N=105) | Hybrid Closed Loop Control (HCL) (N=81) | Predictive Low-Glucose Insulin Suspension (PLGS) (N=79) | Sensor-Augmented Pump (SAP) (N=78)
Chest pain (General disorders) | 0 | 1 | 0 | 1
Hyperglycemia (Blood and lymphatic system disorders) | 3 | 1 | 7 | 4
Fall (General disorders) | 0 | 1 | 4 | 1
Hypoglycemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Gastroenteritis (General disorders) | 0 | 0 | 1 | 0
Wound (General disorders) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 2 | 0
Ketosis (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Foot injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Edema (General disorders) | 0 | 0 | 0 | 1
Abdominal pain (General disorders) | 0 | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Rectal Bleeding (General disorders) | 1 | 0 | 0 | 0
Palpitation (Cardiac disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-05-05): https://cdn.clinicaltrials.gov/large-docs/62/NCT04016662/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-06): https://cdn.clinicaltrials.gov/large-docs/62/NCT04016662/SAP_001.pdf
  • Informed Consent Form (2021-06-03): https://cdn.clinicaltrials.gov/large-docs/62/NCT04016662/ICF_002.pdf